CLINICAL TRIAL: NCT04820257
Title: Home-based Pulmonary Rehabilitation for COPD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marian Papp, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-01151:DNR
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: COPD, Chronic Obstructive Pulmonary Disease
Keywords: tele-health; behavioural change; motivational interviewing; home-based exercise; self-related health; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: starting with a small pilot and will follow with parallell design RCT - starting later
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home based exercise (Experimental): Home based exercise with health coaching
  Interventions: Behavioral: Home based exercise
- Usual care (No Intervention): Usual care, waiting list

INTERVENTIONS:
Behavioral: Home based exercise — Exercise at home and behavioural change to increase daily exercise
  Arms: Home based exercise

SUMMARY:
Objectives The objective of this project is to motivate patients with COPD to incorporate the habit of doing daily mindful physical activity by using the proposed home-based pulmonary rehabilitation program that integrates video guided exercises, activity monitoring daily steps and health coaching. This program will allow patients to complete Pulmonary Rehabilitation (PR) at home and promote behavior change and lead to a more active lifestyle for patients with COPD who have been prescribed PR.

The program will be able to effectively monitor daily step count. A health coach will receive more this detailed data and will guide weekly health coaching sessions designed to increase awareness of the physical activities completed and ignite inner motivation for healthy behaviors.

The proposed PR program is innovative and responds to an unmet need in chronic care for COPD patients in the context of COVID-19 pandemic and it mitigates the common accessibility barriers.

DETAILED DESCRIPTION:
Specific aims will guide the proposed project:

* Aim 1: To determine the feasibility of the proposed home-based PR program. We will additionally address adherence and appropriateness of the program.
* Aim 2: To determine improvements in quality of life and mental health of the proposed home-based PR determined.
* Aim 3: To evaluate if the average number of daily step counts increase after the home-based PR program

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 40 years and older
* FEV1 <80% or less (forced expiratory volume in one second) as documented by pulmonary function.
* Medical diagnosis of COPD, GOLD classification B,D, and C based on symptoms and history of exacerbations.
* The patients must be able to access a smart-phone or computer tablet with internet service.

Exclusion Criteria:

* Unable to perform low intensity exercise.
* Patients with a high likelihood of being lost to follow-up or contact (patients with active chemical dependency), are planning to move, are not living in the healthcare area.
* Patients with an inability to provide good data or follow commands (patients who are disoriented, have a severe neurologic or psychiatric condition).

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Disease specific quality of life | 8-12 weeks
  Chronic Respiratory Questionnaire (CRQ)
Modified Medical Research Council Dyspnea scale (mMRC), | 8-12 weeks
  Dyspnea
COPD assessment Test (CAT) | 8-12 weeks
  assess symptoms of breathing

SECONDARY OUTCOMES:
GAD to asses anxiety and depression symptoms | 8-12 weeks
  assessing anxiety and depression symptoms
Online breathing and mindful movement exercises/ exercise routine | 8-12 weeks
  Total time performing the breathing exercises
Activity monitoring | 8-12 weeks
  number of steps

CONTACTS AND LOCATIONS:
Overall Officials: Marian Papp, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden